CLINICAL TRIAL: NCT00514930
Title: A Multicentre Prospective Clinical Trial of a New Bipolar Radiofrequency Ablation/Aspirator Device (Hexablate) in the Management of Primary and Secondary Liver Cancers
Brief Title: Multicentre Prospective Clinical Trial for RFA Tumour Aspirator Treatment of Primary and Secondary Malignancies of the Liver
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Multicenter hexablate protocol
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Liver Cancer
Keywords: radiofrequency ablation; liver cancer; complications; liver tumors
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

INTERVENTIONS:
Device: Hexablate

SUMMARY:
The primary aim for this trial is to assess whether the RFA aspirator device is safe and of clinical benefit in patients with primary or secondary malignant liver tumours

DETAILED DESCRIPTION:
Patients with unresectable primary or secondary malignancies of the liver have limited treatment options which often only give a small survival benefit. RFA has been demonstrated to be effective in local tumour eradication and to extend patient survival. In this study RFA aspiration will be used to treat unresectable primary or secondary tumours of the liver. RFA will be used to develop a shell of tissue destruction around the tumour, with aspiration removing tissue and fluid from the centre of the lesion. The potential advantages of aspirating during ablation could be to reduce aerosol spread of tumour within the liver parenchyma and peritoneum. Additionally, aspirating the ablated tissue may reduce the incidence of systemic side effects related to RFA when larger lesions are treated. This study would establish the safety and efficiacy of RFA aspiration in the treatment of unresectable primary/secondary malignancies of the liver.

This protocol is for a prospective multi-centre clinical trial of the use of RFA aspiration in the treatment of patients with primary/secondary malignancies of the liver, which are not suitable for formal liver resection. The basis for unresectability being the presence of extra-hepatic disease, limited liver synthetic function, co-morbidity (ASA>3), bilobar disease and anatomical location. Early and late complications relating to the usage of the RFA aspirator will be analysed. Additionally, local recurrence and long term survival will be assessed. If the use of the RFA aspirator produces improved survival with minimal morbidity and mortality. Then these initial results will justify further in depth studies to establish its clinical role.

II. SPECIFIC AIMS/OBJECTIVES

The primary aim for this trial is to assess whether the RFA aspirator device is safe and of clinical benefit in patients with primary or secondary malignant liver tumours.

III. STUDY OVERVIEW

It is anticipated that 100-200 participants will be recruited. The time period for patient recruitment will be for 2 years with follow up for 3 years. The total study period will be 5 years in order to allow the assessment of complications, local ablation success and survival benefit.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 18 years and older.
* Have unresectable primary/secondary malignant tumours of the liver. Unresectable criteria being the presence of extra-hepatic disease, limited liver synthetic function, co-morbidity (ASA 3), bilobar disease and anatomical location.
* Study specific signed informed consent will also have to be completed to allow patient inclusion.

Exclusion Criteria:

* Age younger than 18 years old
* Pregnant women
* Uncorrectable coagulopathy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-02; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
To estimate the local and remote intra-hepatic and extra-hepatic recurrence rates and their impact on survival. | 2 years

SECONDARY OUTCOMES:
Complications and unexpected adverse events (early and late) related to RFA aspirator treatment to be assessed. Data points to be collected as per proforma for trial. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Zacharoulis, M.D., Principal Investigator — University of Thessaly; Nagy Habib, Professor, Study Chair — Imperial College London U.K.; Giuseppe Navarra, Professor, Study Director — University of Messina
Locations (1):
- C. Hatzitheofilou, Larissa, Greece

REFERENCES:
- [Derived] Zacharoulis D, Khorsandi SE, Vavra P, Dostalik J, Navarra G, Nicholls JP, Jiao LR, Habib NA. Pilot study for a new bipolar radiofrequency ablation/aspirator device in the management of primary and secondary liver cancers. Liver Int. 2009 Jul;29(6):824-30. doi: 10.1111/j.1478-3231.2008.01910.x. PMID 19638109